CLINICAL TRIAL: NCT02218151
Title: Patient-Centered Medical Home Care for Hematopoietic Stem Cell Transplantation: A Randomized Phase 2 Study
Brief Title: Medical Home Care for Hematopoietic Stem Cell Transplantation Phase 2
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low accrual due to covid-19 and resulting staffing shortages
Sponsor: Duke University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00051024; R01CA203950-03 (NIH)
Record Dates: First submitted 2014-08-14; First posted 2014-08-15 (Estimated); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Blood Disorders
Keywords: Hematopoietic; Stem Cell; Transplant; patient-centered; Microbiota; GVHD
MeSH Terms: conditions — Hematologic Diseases | interventions — Patient-Centered Care; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Patient-Centered Medical Home (PCMH) (Experimental): Day-to-Day Care:
  Advanced Practice Providers (APP) will travel to subjects' homes in the morning, where they will perform the same daily assessment as standard care. They will draw labs and bring them back to the hospital for processing. When results are available, a second home visit is made to deliver necessary interventions. Subjects will have internet access through cellular-networked iPads and have daily videoconferences with their physicians. Daily follow up at home will continue until discharge as per above criteria.
  Caregivers: identified by the subject as the person taking primary care of them will answer surveys and also collect stool samples to analyze in conjunction with those from subjects.
  Interventions: Other: Patient-Centered Medical Home (PCMH)
- Standard Care (Active Comparator): These subjects will begin as inpatients or outpatients, where advanced practice providers (APPs) (nurse practitioners and physician assistants) will perform histories and physical exams. Nurses will collect labs and providers will enter orders in our electronic health record (EHR). All steps will be repeated daily until discharge to home. Suitability for discharge is determined by standard clinical criteria including stable blood counts, freedom from active or severe complications (e.g. active infection, severe GVHD), and ability to care for self.
  Caregivers: identified by the subject as the person taking primary care of them will answer surveys and also collect stool samples to analyze in conjunction with those from subjects.
  Interventions: Other: Standard Care

INTERVENTIONS:
Other: Patient-Centered Medical Home (PCMH) — Subjects will receive their conditioning chemotherapy +/- radiation and stem cells in the hospital or day hospital, after which they will receive care during the neutropenic/recovery period at home. Advanced Practice Providers (APP) will travel to subjects' homes in the morning, where they will perform the same daily assessment as standard care. They will draw labs and bring them back to the hospital for processing. When results are available, a second home visit is made to deliver necessary interventions. Subjects will have internet access through cellular-networked iPads and have daily videoconferences with their physicians. Daily follow up at home will continue until discharge as per above criteria.
  Arms: Patient-Centered Medical Home (PCMH)
Other: Standard Care — Subjects will receive their conditioning chemotherapy +/- radiation and stem cells in the hospital or day hospital, after which they will receive care during the neutropenic/recovery period inpatient or outpatient. Advanced practice providers (APPs) will perform histories and physical exams. Nurses will collect labs and inpatient rounds occur twice daily, or for outpatients receiving care through our outpatient clinics, a healthcare provider typically sees them daily for the first month following transplant or discharge from the day hospital.
  Arms: Standard Care

SUMMARY:
Hematopoietic stem cell transplantation (HCT) has the potential to cure a variety of malignant and non-malignant diseases. However, it is associated with significant morbidity, and treatment-related mortality. This is due in large part to the prolonged pancytopenia and immunosuppression associated with the preparatory regimen of chemotherapy and/or radiation and the wait until engraftment of the transplanted hematopoietic stem cells. During this vulnerable period, infectious complications are common. Historically HCT patients were kept in protected environments to safeguard their health during the pancytopenic phase; despite these measures, infectious complications and graft versus host disease (GVHD) remained common and lead to significant morbidity and mortality after HCT. Currently patients are still closely watched in the inpatient or day hospital environment, though recent practices allow patients more freedom. This study randomizes eligible patients to receive post-transplant care at home vs. in the hospital or clinic, per standard of care. The primary objective is to compare the incidence of grade II-IV acute GVHD at 6 months in patients receiving patient-centered medical home (PCMH) vs standard care.

DETAILED DESCRIPTION:
The patient-centered medical home (PCMH) is an exciting strategy that has the potential to revolutionize hematopoietic stem cell transplantation (HCT). Traditionally, home care has been used for palliative care in end-stage cancer patients and in geriatrics. More recently the PCMH has gained increasing adoption for both primary care and care of medically complex patients. The core of the PCMH lies in the interaction between the healthcare team, the patient's family and support, and above all, the patient. These interactions can be enhanced through health information technologies such as the electronic health record (EHR) and videoconferencing via iPads. In addition, collection of patient reported outcomes (PRO) will allow feedback and adjustments.

This integration is especially important when considering the multiple complicated needs of the HCT patient: navigating a Byzantine healthcare system that often requires input and coordination from multiple specialists including transplanters, hematologists, infectious disease physicians, gastroenterologists, psychiatrists, nutritionists, pharmacists, social workers, financial coordinators, etc.; managing medication regimens to prevent infections, GVHD, and other complications (not to mention avoiding drug and food interactions); adjusting to multiple side effects including fatigue, weakness, anorexia, nausea, vomiting, diarrhea, rashes, pain, anxiety, stress, organ failure, etc.; the sheer amount of time required for healthcare visits, lab draws, waiting for results, infusions, transfusions, etc.; physical and psychosocial struggles of living with a life-threatening disease; and the burdens of a treatment that often seems as debilitating as the disease. The PCMH provides patient-centered, comprehensive, accessible, and coordinated care and a systems-based approach to quality and safety: these attributes are essential to the successful care of the complicated HCT patient. this approach has the potential to lower overall costs while preserving or increasing the quality of care.

ELIGIBILITY:
Inclusion Criteria:

1. Scheduled to undergo a hematopoietic stem cell transplant for any cancer or non-cancer illness
2. Age 18-80 years of age
3. Karnofsky Performance Scale (KPS)> 80
4. A home that is deemed, upon inspection, in suitable condition to serve as a medical home, within a 90-minute driving distance of Duke

Exclusion Criteria:

1. Lack of a caregiver
2. Pregnant women
3. Patients with a documented active infection prior to starting their preparative regimen. This includes grade 3 or higher viral, bacterial, or fungal infection.
4. Use of homeopathic medications or probiotics that may impact gut microbiota

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2014-09-03 (Actual); Primary Completion 2021-07-12 (Actual); Study Completion 2022-02-14 (Actual)

PRIMARY OUTCOMES:
Acute Graft Versus Host Disease (aGVHD) | 6 months
  The primary endpoint is the incidence (number of events) of grade II-IV acute GVHD at 6 months. GVHD will be evaluated daily by advanced practice providers (APPs) according to standard criteria. The investigators will compare GVHD incidence rates between treatment arms using survival type regression modeling that takes competing risks into account. They will examine cause-specific Cox proportional hazards models as well as the proportional subdistribution hazard regression model developed by Fine and Gray. While the primary treatment comparison will be unadjusted, adjustment for covariates to explore the impact of various risk factors will also be performed.

SECONDARY OUTCOMES:
Rate of Infection | 1 year
  Rates of bacterial, fungal, and viral infections as well as overall infections at one year.
Disease Free Survival (DFS) | 1 year
  Disease free survival at one year.
Overall Survival | 1 year
  Overall survival at one year.

OTHER OUTCOMES:
Comparison of Gut Microbiota | 6 months
  Shannon diversity index will be compared using unpaired two-sided Student's t tests with a more stringent cut-off of 0.0125 given multiple comparisons, by the Bonferroni correction for 4 time periods of independent comparisons. Comparisons of bacterial populations will be made by using the Adonis non-parametric method from within the Qiime package using UnifFrac distance matrices from the populations being compared. P values will be calculated with α= 0.05. Metastatistics will be used for further statistical analyses of population structure, membership, and diversity with metadata such as time from transplant and dietary measurements such as caloric intake. Changes in specific bacterial families of interest will be compared using a two-sided Student's t test, with normality confirmed by D'Agostino and Pearson omnibus test with p≤0.05. All other comparisons will be done using two-sided Mann-Whitney tests.

CONTACTS AND LOCATIONS:
Overall Officials: Nelson J C, MD, MBA, Principal Investigator — Duke University
Locations (1):
- Duke University Adult Bone Marrow Transplant Clinic, Durham, North Carolina, United States